CLINICAL TRIAL: NCT02880371
Title: A Phase 1b/2 Study of ARRY-382 in Combination With Pembrolizumab, a Programmed Cell Death Receptor 1 (PD-1) Antibody, for the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Study of ARRY-382 in Combination With Pembrolizumab for the Treatment of Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was halted prematurely due to insufficient efficacy. Not due to safety reasons.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-382-201; C4261001 (Other: Alias Study Number)
Record Dates: First submitted 2016-08-02; First posted 2016-08-26 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Pembrolizumab; ARRY-382; CSF-1R; CSF1R; cfms
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b/Part A (Experimental): Patients in Part A will receive escalating doses of single-agent ARRY-382 in combination with 2 mg/kg pembrolizumab.
  Interventions: Drug: ARRY-382; Drug: Pembrolizumab
- Phase 2 (Experimental): Patients in Phase 2 will receive the MTD/RP2D dose of ARRY-382 determined during Part A in combination with 200mg pembrolizumab.
  Interventions: Drug: ARRY-382; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ARRY-382 — ARRAY-382 will be taken by mouth once daily at a fixed dose.
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously over 30 minutes every 3 weeks.

SUMMARY:
This is an open-label, multicenter Phase 1b/2 study to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of ARRY-382 in combination with pembrolizumab in adult patients with selected advanced solid tumors (Part A/Phase 1b); and to estimate the efficacy of the combination in three separate cohorts: 1) patients with advanced solid tumors that have progressed on prior PD-1/PD-L1inhibitors, 2) patients with platinum-resistant ovarian cancer and 3) patients with pancreatic ductal adenocarcinoma (Phase 2).

DETAILED DESCRIPTION:
ARRY-382 is an inhibitor of CSF1R (colony-stimulating factor-1 receptor).

Each phase of the study consists of a 28-day screening period; 21-day treatment cycles with the combination of ARRY-382 and pembrolizumab until disease progression as determined by the Investigator, unacceptable toxicity, withdrawal of consent, or death (or other discontinuation criteria are met), and a 30-day safety follow-up period. Patients in all cohorts/phases will be monitored for overall survival (OS) until 1 year after the date of the last patient's first visit.

ELIGIBILITY:
Key Inclusion Criteria

All Study Parts:

* Diagnosis of cancer that has been histologically or cytologically confirmed
* Eastern Cooperative Oncology Group Performance Status of 0 or 1

Part A (1 of the following):

* Ovarian cancer, triple-negative breast cancer, head and neck squamous cell cancer, bladder cancer, metastatic colorectal cancer, pancreatic ductal adenocarcinoma, or gastric cancer that is measurable or evaluable, nonmeasurable as defined by RECIST v1.1 and meets 1 of the following criteria:

  * is refractory to standard of care
  * no standard therapy available
  * patient refuses standard therapy
* Advanced, unresectable, or metastatic melanoma with or without prior treatment and measurable or evaluable, nonmeasurable disease as defined by RECIST v1.1
* Advanced/metastatic PD-L1-positive NSCLC (defined as a tumor proportion score [TPS] ≥ 50%) with measurable or evaluable, non-measurable disease as defined by RECIST v1.1 (1 of the following):

  * 1) No prior systemic chemotherapy if tumor does not have EGFR or ALK genomic aberrations
  * 2) Disease progression on or after platinum-containing chemotherapy;
  * 3) If tumor has EGFR or ALK genomic aberrations, disease progression on an FDA-approved therapy for EGFR or ALK genomic tumor aberrations

Phase 2 (1 of the following):

* Advanced/metastatic solid tumor with PD as defined by RECIST 1.1 or irRC on an anti-PD-1- or anti-PD-L1-containing regimen as their most recent prior therapy
* Advanced/metastatic epithelial ovarian cancer, peritoneal cancer or tubal cancer with measurable disease as defined by RECIST 1.1, that had progressed within 6 months of completing ≥ 4 cycles of platinum-based therapy
* Advanced/metastatic PDA that is locally advanced, unresectable or metastatic with measurable disease as defined by RECIST v1.1 in patients who have received at least one prior line of systemic therapy for their disease

Key Exclusion Criteria

1. Prior treatment as follows:

   * Part A: an immune CPI (e.g., PD-1, PD-L1, or cytotoxic T-lymphocyte antigen 4 [CTLA-4] inhibitor).

   NOTE: For patients with melanoma, prior treatment with ipilimumab is allowed if it was administered as adjuvant therapy and treatment was completed at least 3 months prior to enrollment.
   * Phase 2:

     * A CSF-1R inhibitor or CSF-1 (or MCSF) inhibitor.
     * prOVCA and PDA patients only: an immune CPI (e.g., PD-1, PD-L1, or CTLA-4 inhibitor)
2. Symptomatic brain metastasis at screening
3. Active autoimmune disease, documented history of autoimmune syndrome or disease, or a chronic medical condition that requires chronic steroid therapy or immunosuppressive medication
4. History of pneumonitis or interstitial lung disease
5. Severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient an inappropriate candidate for the study
6. Ocular melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (30):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Hem-Onc Associates of Treasure Coast, Port Saint Lucie, Florida
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - PPG, Fort Wayne, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Hall-Perrine Cancer Center Laboratory, Cedar Rapids, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Labs - Rochester Superior, Rochester, Minnesota
  - Regions Cancer Care Center, Saint Paul, Minnesota
  - Regions Hospital Pharmacy, Saint Paul, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - HealthPartners Neurosciences Center, Saint Paul, Minnesota
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Health Cancer Center, San Antonio, Texas
  - UTAH Cancer Specialists, Salt Lake City, Utah
  - ARUP Laboratories, Inc., Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - UVA Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Johnson M, Dudek AZ, Sukari A, Call J, Kunk PR, Lewis K, Gainor JF, Sarantopoulos J, Lee P, Golden A, Harney A, Rothenberg SM, Zhang Y, Goldman JW. ARRY-382 in Combination with Pembrolizumab in Patients with Advanced Solid Tumors: Results from a Phase 1b/2 Study. Clin Cancer Res. 2022 Jun 13;28(12):2517-2526. doi: 10.1158/1078-0432.CCR-21-3009. PMID 35302585
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-382-201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 phases: Phase 1B and 2. Originally, Phase 1b of the study had Part A and B. Part A was dose escalation in participants with selected advanced solid tumors. Part B was expansion in melanoma participants. Part C was a part of Phase 2, in participants with non-small cell lung cancer (NSCLC).
Pre-assignment Details: There was an amendment in protocol, which removed originally designed Part B and C, due to low enrolment. Post-implementation of this amendment 2, Part B and C were replaced with 3 cohorts in Phase 2. Study then had Part A (Phase 1b), and 3 cohorts in Phase 2. Cohorts of Phase 2 were as follows: 1) PD-1/PD-L1 inhibitor-refractory cohort, 2) pancreatic ductal adenocarcinoma cohort and 3) platinum-resistant ovarian cancer cohort.
Groups:
- Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab: Participants with selected advanced solid tumors received ARRY-382 capsules at a dose of 200 milligrams (mg) orally, once daily (QD) in combination with pembrolizumab at a dose of 2 milligram per kilogram (mg/kg) intravenously (IV) every 3 weeks (Q3W) in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab: Participants with selected advanced solid tumors received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 2 mg/kg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab: Participants with selected advanced solid tumors received ARRY-382 capsules at a dose of 400 mg orally, QD in combination with pembrolizumab at a dose of 2 mg/kg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 1b, Part B: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab: Participants with melanoma received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 2 mg/kg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 2, Part C: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab: Participants with NSCLC received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 2 mg/kg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort: Participants who progressed on a programmed cell death receptor 1 (PD-1)/ programmed cell death ligand 1 (PD-L1) inhibitor-containing regimen as their most recent prior line of therapy and were new to prior colony-stimulating factor 1 receptor (CSF-1R) or colony-stimulating factor 1(CSF-1) inhibitors were included in this reporting arm. Participants received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 200 mg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort: Participants with PDA who had at least 1 prior line of therapy and were new to prior checkpoint inhibitor (CPI) therapy and to prior CSF-1R or CSF-1 inhibitors were included in this reporting arm. Participants received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 200 mg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort: Participants with prOVCA who had at least 1 prior line of therapy and were new to prior CPI therapy and to prior CSF-1R or CSF-1 inhibitors were included in this reporting arm. Participants received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 200 mg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
Period: Phase 1b
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part B: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2, Part C: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Started | 6 | 7 | 7 | 1 | 0 | 0 | 0 | 0
Treated | 6 | 6 | 7 | 1 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 7 | 6 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participants terminated by Sponsor | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 4 | 6 | 5 | 1 | 0 | 0 | 0 | 0
Not completed — Enrolled but not Treated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part B: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2, Part C: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Started | 0 (Participants of Phase 1b were different from Phase 2.) | 0 (Participants of Phase 1b were different from Phase 2.) | 0 (Participants of Phase 1b were different from Phase 2.) | 0 (Participants of Phase 1b were different from Phase 2.) | 2 (Participants enrolled for Phase 2 were different from participants enrolled for Phase 1b.) | 20 (Participants enrolled for Phase 2 were different from participants enrolled for Phase 1b.) | 28 (Participants enrolled for Phase 2 were different from participants enrolled for Phase 1b.) | 11 (Participants enrolled for Phase 2 were different from participants enrolled for Phase 1b.)
Treated | 0 | 0 | 0 | 0 | 2 | 19 | 27 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 20 | 28 | 11
Not completed — Enrolled but not Treated | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Participants terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 6 | 1 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 10 | 20 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — End of Study page not completed by error | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported for full analysis set (FAS). FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Groups:
- Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab: Participants with selected advanced solid tumors received ARRY-382 capsules at a dose of 200 mg orally, QD in combination with pembrolizumab at a dose of 2 mg/kg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort: Participants who progressed on a PD-1/ PD-L1 inhibitor-containing regimen as their most recent prior line of therapy and were new to prior CSF-1R or CSF-1 inhibitors were included in this reporting arm. Participants received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 200 mg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort: Participants with PDA who had at least 1 prior line of therapy and were new to prior CPI therapy and to prior CSF-1R or CSF-1 inhibitors were included in this reporting arm. Participants received ARRY-382 capsules at a dose of 300 mg orally, QD in combination with pembrolizumab at a dose of 200 mg IV Q3W in each 21-day treatment cycle until disease progression, participant refusal, lost to follow-up, unacceptable toxicity, or the study termination by the sponsor and a 30-day safety follow-up period.
- Total: Total of all reporting groups
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part B: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2, Part C: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort | Total
Number analyzed (Participants) | 6 | 6 | 7 | 1 | 2 | 19 | 27 | 11 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (12.4) | 52.2 (16.0) | 54.7 (12.9) | 68.0 (NA) — Since only 1 evaluable participant, standard deviation could not be calculated. | 47.0 (0.0) | 63.1 (12.0) | 65.0 (9.6) | 59.3 (13.1) | 61.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 0 | 0 | 12 | 12 | 11 | 44
  Male | 4 | 3 | 3 | 1 | 2 | 7 | 15 | 0 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 6 | 7 | 1 | 2 | 18 | 23 | 10 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 5
  White | 5 | 6 | 7 | 1 | 2 | 15 | 23 | 9 | 68
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b, Part A: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT: adverse event (AE) or abnormal laboratory value not clearly attributable to an extraneous cause, such as disease progression, intercurrent illness, or concomitant medications occurring during 21 days of Cycle 1, met 1 of the criteria A) nonhematologic AEs: recurring grade 2 pneumonitis, grade 3 events (irAE, QTcF prolongation, rash; other grade 3/4 except alopecia, nausea, diarrhea, vomiting, tumor flare, pseudoprogression, endocrinopathy); B) hematology AEs/laboratory abnormalities: grade 4 events except lymphopenia, neutropenia, electrolyte imbalances or abnormalities, grade 3 thrombocytopenia, febrile neutropenia, grade 4 AST/ALT elevation, grade 3 AST/ALT elevation lasting >7 days, associated with bilirubin levels>=2*ULN or international normalized ratio >1.5, grade 3 bilirubin elevation >=3, CK elevation >=grade 3 lasting, increase in creatinine >=1.5*baseline value, dose delay (dose interruption for >14 days) or other (inability to receive at least 67% of ARRY-382 doses).
Time Frame: Cycle 1 (up to 21 days)
Population: Dose-determining set (DDS) included all participants in Phase 1b who received at least 67% of the planned cumulative dose of ARRY-382 during Cycle 1 or discontinued the treatment because of DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab
Number analyzed (Participants) | 6 | 6 | 7
Participants | 0 | 1 | 2

2. Primary Outcome: Phase 2 Cohorts: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator review of radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. As per RECIST v1.1: CR = disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures less than (<) 10 millimeter (mm). PR = at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. Non-target lesions must be non-progressive disease (PD). The analysis was based on confirmed responses for which CR or PR must be confirmed by repeat disease assessment studies performed no less than 4 weeks after the criteria for response were first met to qualify as CR or PR, respectively.
Time Frame: From day of first dose to 30 days after last dose (maximum up to 13.5 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 19 | 27 | 11
percentage of participants | 0.0 [0.0 to 17.6] | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 28.5]

3. Secondary Outcome: Phase 1b, Part A: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a BOR of CR or PR as determined by investigator review of radiographic disease assessments per RECIST v1.1. As per RECIST v1.1: CR = disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. PR = at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. Non-target lesions must be non-PD. The analysis was based on confirmed responses for which CR or PR must be confirmed by repeat disease assessment studies performed no less than 4 weeks after the criteria for response were first met to qualify as CR or PR, respectively.
Time Frame: From day of first dose to 30 days after last dose (maximum up to 34.7 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab
Number analyzed (Participants) | 6 | 6 | 7
percentage of participants | 16.7 [0.4 to 64.1] | 16.7 [0.0 to 64.1] | 0.0 [0.0 to 41.0]

4. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Duration of Response (DOR)
Description: DOR was defined as the time from the date of the first documented response (CR or PR) to the earliest date of disease progression, or death due to any cause after achieving a response. As per RECIST v1.1: CR = disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures < 10 mm. PR = at least a 30% decrease in the sum of measures (longest diameter for tumor lesions and short axis measure for nodes) of target lesions, taking as reference the baseline sum of diameters. PD = at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >= 5 mm or appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions. DOR was estimated using the Kaplan-Meier method.
Time Frame: From date of first documented CR or PR up to disease progression or death (for Phase 1b: maximum up to 34.7 months, for Phase 2: maximum up to 13.5 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab. This outcome measure was evaluated in participants who achieved an objective response. "Overall Number of participants Analyzed" =0, signifies participants did not had documented CR or PR for respective reporting arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 1 | 1 | 0 | 0 | 1 | 0
months | 29.2 [NA to NA] — Upper and lower limit of confidence interval (CI) not reached due to less number of participants with events. | 3.1 [NA to NA] — Upper and lower limit of CI not reached due to less number of participants with events. |  |  | 2.4 [NA to NA] — Upper and lower limit of CI not reached due to less number of participants with events. |

5. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study drug to the earliest date of disease progression per RECIST v1.1, or death due to any cause, whichever occurs first. If a participant did not have a PFS event at the time of the analysis cut-off or at the start of any new anticancer therapy, PFS was censored at the date of last adequate tumor assessment. PD = at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >= 5 mm or appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions.
Time Frame: From day of first dose until disease progression or death due to any cause or till last tumor assessment date (for Phase 1b: maximum up to 34.7 months, for Phase 2: maximum up to 13.5 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
months | 4.7 [1.4 to 33.1] | 2.3 [1.3 to 5.7] | 1.4 [0.5 to 2.6] | 1.6 [1.3 to 4.4] | 1.4 [0.9 to 2.8] | 2.1 [1.2 to 4.1]

6. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Overall Survival (OS)
Description: OS was defined as the time from the start of treatment to the date of death due to any cause. If a death was not observed by the date of the analysis cut-off, OS was censored at the date of last contact. OS was estimated using the Kaplan-Meier method.
Time Frame: From day of first dose till death due to any cause or date of last contact (for Phase 1b: maximum up to 34.7 months, for Phase 2: maximum up to 13.5 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
months | 14.7 [5.2 to NA] — Upper limit of CI not reached due to less number of participants with events. | 7.4 [2.1 to 14.1] | 6.5 [1.0 to NA] — Upper limit of CI not reached due to less number of participants with events. | 12.4 [3.6 to NA] — Upper limit of CI not reached due to less number of participants with events. | 2.2 [1.5 to 4.9] | NA [5.3 to NA] — Median and upper limit of CI not reached due to less number of participants with events.

7. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Percentage of Participants With Immune-Related Response Rate (irRR)
Description: irRR was defined as the percentage of participants who achieved immune-related best overall response (irBOR) of immune-related CR (irCR) or immune-related PR (irPR), as determined by the investigator per immune related response criteria (irRC). irBOR was the best response using irRC recorded from the start of study treatment until the end of treatment. irCR was the disappearance of all target lesions, irPR was a decrease in tumor burden by 50% or greater by a consecutive assessment at least 4 weeks after first documentation.
Time Frame: From day of first dose till up to end of study treatment (for Phase 1b: maximum up to 33.7 months, for Phase 2: maximum up to 12.5 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
percentage of participants | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 17.6] | 3.7 [0.1 to 19.0] | 0.0 [0.0 to 28.5]

8. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Immune-Related Progression-Free Survival (irPFS)
Description: irPFS was defined as the time from the start of treatment to the time of first documented progression per irRC, or death due to any cause. irRC criteria for progression for 1) Measurable new lesions: incorporated into the tumor burden (eg, added to the index lesions); do not define progression unless the total measurable tumor burden increases by the required amount (25%); 2) New non-measurable lesions: not considered progression if the total measurable tumor burden is stable or shrinking. For the analysis of irPFS, Kaplan-Meier method was used.
Time Frame: From the start of treatment to the time of first documented progression, or death (for Phase 1b: maximum up to 34.7 months, for Phase 2: maximum up to 13.5 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
months | 3.0 [1.4 to 16.1] | 2.5 [1.4 to 7.1] | 1.3 [0.5 to 1.5] | 1.5 [1.3 to 4.3] | 1.3 [0.9 to 2.7] | 2.5 [1.2 to NA] — Upper limit of CI not reached due to less number of participants with events.

9. Secondary Outcome: Phase 2 prOVCA: Change From Baseline in Tumor Markers at Day 1 of Cycle 1, 2, 3, 4, 5, 6, 7, Day 8, 15 of Cycle 1 and Treatment Discontinuation
Description: Tumor markers were measured for tumor type from serum samples obtained from participants in Phase 2. Mean change from baseline was reported in this outcome measure.
Time Frame: Baseline, Day 1 of Cycle 1, 2, 3, 4, 5, 6, 7, Day 8, 15 of Cycle 1 and Treatment discontinuation (before 13.5 months)
Population: FAS included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab. This outcome measure was planned in prOVCA cohort. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 11
microgram per milliliter
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 578.6 (626.3302643)
  Cycle 1 Day 8 | 803.3181818 (808.9155788)
  Cycle 1 Day 15: number analyzed (Participants) | 9
  Cycle 1 Day 15 | 1279.833333 (1298.144638)
  Cycle 2 Day 1: number analyzed (Participants) | 10
  Cycle 2 Day 1 | 1485.6 (1368.310653)
  Cycle 3 Day 1: number analyzed (Participants) | 5
  Cycle 3 Day 1 | 1558.4 (1502.22728)
  Cycle 4 Day 1: number analyzed (Participants) | 1
  Cycle 4 Day 1 | 1980 (NA) — Since only 1 evaluable participant, standard deviation could not be calculated.
  Cycle 5 Day 1: number analyzed (Participants) | 1
  Cycle 5 Day 1 | 778 (NA) — Since only 1 evaluable participant, standard deviation could not be calculated.
  Cycle 6 Day 1: number analyzed (Participants) | 1
  Cycle 6 Day 1 | 1730 (NA) — Since only 1 evaluable participant, standard deviation could not be calculated.
  Cycle 7 Day 1: number analyzed (Participants) | 1
  Cycle 7 Day 1 | 2080 (NA) — Since only 1 evaluable participant, standard deviation could not be calculated.
  Treatment discontinuation: number analyzed (Participants) | 6
  Treatment discontinuation | 1743.833333 (1817.18193)

10. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: First dose of study drug up to 30 days after last dose (for Phase 1b: maximum up to 34.7 months, for Phase 2: maximum up to 13.5 months)
Population: Safety set included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
Participants
  AEs | 6 | 6 | 6 | 19 | 27 | 10
  SAEs | 3 | 1 | 3 | 8 | 15 | 5

11. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Number of Participants With Newly Occurring or Worsening Serum Chemistry Laboratory Abnormalities Graded by Common Terminology Criteria for Adverse Events (CTCAE) Grade 4.03
Description: Abnormalities: Albumin (hypoalbuminemia),Alkaline phosphatase (ALP increased), Alanine aminotransferase (ALT increased), Aspartate aminotransferase (AST increased),Total bilirubin (TBL increased), Creatinine (increased), Corrected calcium (hypocalcemia/hypercalcemia), Creatine kinase (CK increased), Glucose (hypoglycemia/hyperglycemia), Amylase (increased), Lipase (increased) ,Phosphate (hypophosphatemia), Magnesium (hypomagnesemia/hypermagnesemia), Potassium (hypokalemia/hyperkalemia), Sodium (hyponatremia/hypernatremia). Participants with all grades and grade 3/4 abnormalities were reported. Test abnormalities were graded by CTCAE v4.03 as Grade 1=mild; Grade 2=moderate; Grade 3/Grade 4=severe/life-threatening.
Time Frame: as for outcome 10
Population: Safety set included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
Participants
  Albumin (grams per liter [g/L]), Hypo: All Grades | 4 | 2 | 4 | 5 | 10 | 2
  Albumin (g/L), Hypo: Grade 3/4 | 1 | 0 | 1 | 0 | 3 | 0
  Alkaline Phosphatase (units per liter [U/L]), Hyper: All Grades | 5 | 3 | 4 | 11 | 17 | 6
  Alkaline Phosphatase (U/L), Hyper: Grade 3/4 | 1 | 0 | 0 | 0 | 4 | 0
  Alanine Aminotransferase (U/L), Hyper: All Grades | 2 | 3 | 4 | 8 | 12 | 7
  Alanine Aminotransferase (U/L), Hyper: Grade 3/4 | 0 | 1 | 1 | 2 | 1 | 3
  Amylase (U/L), Hyper: All Grades | 3 | 4 | 2 | 11 | 7 | 7
  Amylase (U/L), Hyper: Grade 3/4 | 2 | 0 | 0 | 3 | 1 | 1
  Aspartate Aminotransferase (U/L), Hyper: All Grades | 5 | 6 | 6 | 17 | 23 | 11
  Aspartate Aminotransferase (U/L), Hyper: Grade 3/4 | 1 | 2 | 2 | 4 | 5 | 2
  Bilirubin (micromoles per liter [umol/L]), Hyper: All Grades | 1 | 0 | 1 | 3 | 7 | 1
  Bilirubin (umol/L), Hyper: Grade 3/4 | 0 | 0 | 1 | 0 | 3 | 0
  Calcium (millimoles per liter [mmol/L]), Hypo: All Grades | 1 | 1 | 1 | 1 | 0 | 2
  Calcium (mmol/L), Hypo: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium (mmol/L), Hyper: All Grades | 0 | 0 | 0 | 1 | 1 | 0
  Calcium (mmol/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase (U/L), Hyper: All Grades | 5 | 5 | 5 | 16 | 20 | 7
  Creatine Kinase (U/L), Hyper: Grade 3/4 | 0 | 2 | 1 | 3 | 2 | 2
  Creatinine (umol/L), Hyper: All Grades | 2 | 2 | 1 | 7 | 6 | 2
  Creatinine (umol/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 1 | 0 | 0
  Glucose (mmol/L), Hypo: All Grades | 0 | 1 | 0 | 3 | 1 | 0
  Glucose (mmol/L), Hypo: Grade 3/4 | 0 | 0 | 0 | 1 | 0 | 0
  Glucose (mmol/L), Hyper: All Grades | 1 | 1 | 1 | 0 | 0 | 2
  Glucose (mmol/L), Hyper: Grade 3/4 | 1 | 1 | 1 | 0 | 0 | 2
  Potassium (mmol/L), Hypo: All Grades | 1 | 2 | 3 | 7 | 6 | 4
  Potassium (mmol/L), Hypo: Grade 3/4 | 1 | 0 | 0 | 2 | 1 | 0
  Potassium (mmol/L), Hyper: All Grades | 0 | 0 | 0 | 1 | 4 | 1
  Potassium (mmol/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase (U/L), Hyper: All Grades | 5 | 4 | 3 | 8 | 2 | 5
  Lipase (U/L), Hyper: Grade 3/4 | 2 | 2 | 0 | 7 | 0 | 2
  Magnesium (mmol/L), Hypo: All Grades | 0 | 1 | 0 | 5 | 4 | 3
  Magnesium (mmol/L), Hypo: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Magnesium (mmol/L), Hyper: All Grades | 2 | 1 | 2 | 3 | 5 | 0
  Magnesium (mmol/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphate (mmol/L), Hypo: All Grades | 1 | 3 | 0 | 6 | 7 | 2
  Phosphate (mmol/L), Hypo: Grade 3/4 | 1 | 0 | 0 | 2 | 2 | 0
  Sodium (mmol/L), Hypo: All Grades | 3 | 2 | 3 | 8 | 13 | 6
  Sodium (mmol/L), Hypo: Grade 3/4 | 0 | 0 | 1 | 0 | 5 | 1
  Sodium (mmol/L), Hyper: All Grades | 3 | 0 | 0 | 4 | 0 | 0
  Sodium (mmol/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Number of Participants With Newly Occurring or Worsening Hematology and Coagulation Laboratory Abnormalities Graded by CTCAE Grade 4.03
Description: Hematology abnormalities: Hemoglobin (anemia/hemoglobin increased), Platelets (count decreased), Leukocytes (count decreased/increased), Neutrophils (count decreased), Lymphocytes (count increased/decreased). Coagulation abnormalities: International Normalized Ratio (INR increased), Partial thromboplastin time(PTT)/Activated partial thromboplastin Time (aPTT, time prolonged). Abnormalities were graded by CTCAE grade 4.03 as Grade 1= mild; Grade 2 = moderate; Grade 3/Grade 4 = severe/life-threatening. Participants with all grades and grade 3/4 abnormalities were reported.
Time Frame: as for outcome 10
Population: Safety set included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
Participants
  Hemoglobin (g/L), Hypo: All Grades | 3 | 4 | 5 | 12 | 9 | 7
  Hemoglobin (g/L), Hypo: Grade 3/4 | 1 | 0 | 1 | 4 | 2 | 2
  Hemoglobin (g/L), Hyper: All Grades | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin (g/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (10^9/L), Hypo: All Grades | 2 | 1 | 3 | 11 | 11 | 5
  Lymphocytes (10^9/L), Hypo: Grade 3/4 | 2 | 1 | 2 | 5 | 1 | 2
  Lymphocytes (10^9/L), Hyper: All Grades | 0 | 0 | 0 | 0 | 1 | 0
  Lymphocytes (10^9/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (10^9/L), Hypo: All Grades | 1 | 3 | 0 | 1 | 0 | 1
  Neutrophils (10^9/L), Hypo: Grade 3/4 | 1 | 0 | 0 | 1 | 0 | 0
  Platelets (10^9/L), Hypo: All Grades | 1 | 1 | 2 | 2 | 2 | 1
  Platelets (10^9/L), Hypo: Grade 3/4 | 0 | 0 | 0 | 1 | 0 | 0
  Leukocytes (10^9/L), Hypo: All Grades | 2 | 1 | 3 | 4 | 2 | 2
  Leukocytes (10^9/L), Hypo: Grade 3/4 | 1 | 0 | 0 | 1 | 0 | 0
  Leukocytes (10^9/L), Hyper: All Grades | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes (10^9/L), Hyper: Grade 3/4 | 0 | 0 | 0 | 0 | 0 | 0
  Activated Partial Thromboplastin Time (sec), Hyper: All Grades | 2 | 2 | 2 | 6 | 7 | 3
  Activated Partial Thromboplastin Time (sec), Hyper: Grade 3/4 | 0 | 0 | 1 | 2 | 2 | 0
  Prothrombin Intl. Normalized Ratio (INR Units), Hyper: All Grades | 1 | 3 | 2 | 9 | 15 | 3
  Prothrombin Intl. Normalized Ratio (INR Units), Hyper: Grade 3/4 | 0 | 0 | 0 | 2 | 1 | 0

13. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Number of Participants With Newly Occurring Abnormal Liver Function Tests
Description: Liver function parameters/abnormalities: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT): >3* upper limit of normal (ULN), >5*ULN, >8*ULN, >10*ULN, >20*ULN; Bilirubin >1.5*ULN, >2*ULN; Alkaline phosphatase (ALP) >2*ULN, >3*ULN.
Time Frame: as for outcome 10
Population: Safety set included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
Participants
  Alanine Aminotransferase: >3*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Alanine Aminotransferase: >3*ULN | 0 | 2 | 2 | 3 | 2 | 4
  Alanine Aminotransferase: >5*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Alanine Aminotransferase: >5*ULN | 0 | 1 | 1 | 2 | 1 | 3
  Alanine Aminotransferase: >8*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Alanine Aminotransferase: >8*ULN | 0 | 0 | 1 | 2 | 1 | 3
  Alanine Aminotransferase: >10*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Alanine Aminotransferase: >10*ULN | 0 | 0 | 1 | 1 | 1 | 3
  Alanine Aminotransferase: >20*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Alanine Aminotransferase: >20*ULN | 0 | 0 | 0 | 0 | 0 | 1
  Alkaline Phosphatase: >2*ULN: number analyzed (Participants) | 4 | 6 | 5 | 18 | 21 | 11
  Alkaline Phosphatase: >2*ULN | 1 | 3 | 2 | 5 | 12 | 3
  Alkaline Phosphatase: >3*ULN: number analyzed (Participants) | 5 | 6 | 5 | 19 | 25 | 11
  Alkaline Phosphatase: >3*ULN | 1 | 0 | 1 | 4 | 9 | 1
  Aspartate Aminotransferase: >3*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Aspartate Aminotransferase: >3*ULN | 2 | 3 | 4 | 7 | 13 | 5
  Aspartate Aminotransferase: >5*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Aspartate Aminotransferase: >5*ULN | 1 | 2 | 2 | 4 | 5 | 2
  Aspartate Aminotransferase: >8*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Aspartate Aminotransferase: >8*ULN | 0 | 1 | 1 | 1 | 1 | 2
  Aspartate Aminotransferase: >10*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Aspartate Aminotransferase: >10*ULN | 0 | 1 | 1 | 1 | 1 | 2
  Aspartate Aminotransferase: >20*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Aspartate Aminotransferase: >20*ULN | 0 | 0 | 0 | 1 | 0 | 1
  Bilirubin: >1.5*ULN: number analyzed (Participants) | 6 | 6 | 5 | 19 | 25 | 11
  Bilirubin: >1.5*ULN | 0 | 0 | 1 | 1 | 5 | 0
  Bilirubin: >2*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  Bilirubin: >2*ULN | 0 | 0 | 1 | 1 | 4 | 0
  ALT or AST: AT >3*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST: AT >3*ULN | 2 | 3 | 4 | 7 | 13 | 5
  ALT or AST: AT >5*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST: AT >5*ULN | 1 | 2 | 2 | 4 | 5 | 3
  ALT or AST: AT >8*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST: AT >8*ULN | 0 | 1 | 1 | 2 | 1 | 3
  ALT or AST: AT >10*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST: AT >10*ULN | 0 | 1 | 1 | 1 | 1 | 3
  ALT or AST: AT >20*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST: AT >20*ULN | 0 | 0 | 0 | 1 | 0 | 1
  ALT or AST and Total Bilirubin >2*ULN: AT >3*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST and Total Bilirubin >2*ULN: AT >3*ULN | 0 | 0 | 1 | 1 | 4 | 0
  ALT or AST and Total Bilirubin >2*ULN: AT >5*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST and Total Bilirubin >2*ULN: AT >5*ULN | 0 | 0 | 1 | 1 | 0 | 0
  ALT or AST and Total Bilirubin >2*ULN: AT >10*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST and Total Bilirubin >2*ULN: AT >10*ULN | 0 | 0 | 1 | 1 | 0 | 0
  ALP >3*ULN and Total Bilirubin >2*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALP >3*ULN and Total Bilirubin >2*ULN | 0 | 0 | 1 | 1 | 3 | 0
  ALT or AST >3*ULN and ALP <2*ULN and Total Bilirubin >2*ULN: number analyzed (Participants) | 6 | 6 | 6 | 19 | 25 | 11
  ALT or AST >3*ULN and ALP <2*ULN and Total Bilirubin >2*ULN | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Number of Participants With Shift in Thyroid Panel Severity From Baseline Grade to Post Baseline Grades
Description: Thyroid panel laboratory parameters/abnormalities: thyrotropin, free triiodothyronine (T3), free thyroxine (T4). Shift in thyroid panel severity from baseline grade low, normal, high and missing to the post baseline grades as low, normal, high and missing is reported in this outcome measure.
Time Frame: Baseline, 30 days after last dose (for Phase 1b: maximum up to 34.7 months, for Phase 2: maximum up to 13.5 months)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
Participants
  Triiodothyronine, Free: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 2 | 1 | 2 | 6 | 9 | 4
  Triiodothyronine, Free: Low (at baseline) to Low (at post baseline) | 0 | 1 | 1 | 3 | 3 | 4
  Triiodothyronine, Free: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 2 | 1 | 2 | 6 | 9 | 4
  Triiodothyronine, Free: Low (at baseline) to Normal (at post baseline) | 1 | 0 | 0 | 3 | 3 | 0
  Triiodothyronine, Free: Low (at baseline) to High (at post baseline): number analyzed (Participants) | 2 | 1 | 2 | 6 | 9 | 4
  Triiodothyronine, Free: Low (at baseline) to High (at post baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Triiodothyronine, Free: Low (at baseline) to Missing (at post baseline): number analyzed (Participants) | 2 | 1 | 2 | 6 | 9 | 4
  Triiodothyronine, Free: Low (at baseline) to Missing (at post baseline) | 1 | 0 | 1 | 0 | 3 | 0
  Triiodothyronine, Free: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 4 | 4 | 5 | 13 | 18 | 7
  Triiodothyronine, Free: Normal (at baseline) to Low (at post baseline) | 1 | 0 | 2 | 0 | 4 | 0
  Triiodothyronine, Free: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 4 | 4 | 5 | 13 | 18 | 7
  Triiodothyronine, Free: Normal (at baseline) to Normal (at post baseline) | 3 | 2 | 3 | 12 | 12 | 7
  Triiodothyronine, Free: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 4 | 4 | 5 | 13 | 18 | 7
  Triiodothyronine, Free: Normal (at baseline) to High (at post baseline) | 0 | 2 | 0 | 1 | 0 | 0
  Triiodothyronine, Free: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 4 | 4 | 5 | 13 | 18 | 7
  Triiodothyronine, Free: Normal (at baseline) to Missing (at post baseline) | 0 | 0 | 0 | 0 | 2 | 0
  Triiodothyronine, Free: High (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Triiodothyronine, Free: High (at baseline) to Low (at post baseline) |  | 0 |  |  |  |
  Triiodothyronine, Free: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Triiodothyronine, Free: High (at baseline) to Normal (at post baseline) |  | 1 |  |  |  |
  Triiodothyronine, Free: High (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Triiodothyronine, Free: High (at baseline) to High (at post baseline) |  | 0 |  |  |  |
  Triiodothyronine, Free: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Triiodothyronine, Free: High (at baseline) to Missing (at post baseline) |  | 0 |  |  |  |
  Thyroxine, Free: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0
  Thyroxine, Free: Low (at baseline) to Low (at post baseline) |  |  |  | 0 | 2 |
  Thyroxine, Free: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0
  Thyroxine, Free: Low (at baseline) to Normal (at post baseline) |  |  |  | 1 | 0 |
  Thyroxine, Free: Low (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0
  Thyroxine, Free: Low (at baseline) to High (at post baseline) |  |  |  | 0 | 0 |
  Thyroxine, Free: Low (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0
  Thyroxine, Free: Low (at baseline) to Missing (at post baseline) |  |  |  | 0 | 1 |
  Thyroxine, Free: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 5 | 5 | 7 | 15 | 22 | 10
  Thyroxine, Free: Normal (at baseline) to Low (at post baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Thyroxine, Free: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 5 | 5 | 7 | 15 | 22 | 10
  Thyroxine, Free: Normal (at baseline) to Normal (at post baseline) | 3 | 2 | 6 | 12 | 18 | 8
  Thyroxine, Free: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 5 | 5 | 7 | 15 | 22 | 10
  Thyroxine, Free: Normal (at baseline) to High (at post baseline) | 1 | 3 | 0 | 3 | 0 | 2
  Thyroxine, Free: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 5 | 5 | 7 | 15 | 22 | 10
  Thyroxine, Free: Normal (at baseline) to Missing (at post baseline) | 1 | 0 | 1 | 0 | 4 | 0
  Thyroxine, Free: High (at baseline) to Low (at post baseline): number analyzed (Participants) | 1 | 1 | 0 | 3 | 2 | 1
  Thyroxine, Free: High (at baseline) to Low (at post baseline) | 0 | 0 |  | 0 | 0 | 0
  Thyroxine, Free: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 1 | 1 | 0 | 3 | 2 | 1
  Thyroxine, Free: High (at baseline) to Normal (at post baseline) | 0 | 0 |  | 1 | 0 | 0
  Thyroxine, Free: High (at baseline) to High (at post baseline): number analyzed (Participants) | 1 | 1 | 0 | 3 | 2 | 1
  Thyroxine, Free: High (at baseline) to High (at post baseline) | 1 | 1 |  | 2 | 2 | 1
  Thyroxine, Free: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 1 | 1 | 0 | 3 | 2 | 1
  Thyroxine, Free: High (at baseline) to Missing (at post baseline) | 0 | 0 |  | 0 | 0 | 0
  Thyrotropin: Low (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Thyrotropin: Low (at baseline) to Low (at post baseline) |  | 0 |  |  |  |
  Thyrotropin: Low (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Thyrotropin: Low (at baseline) to Normal (at post baseline) |  | 1 |  |  |  |
  Thyrotropin: Low (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Thyrotropin: Low (at baseline) to High (at post baseline) |  | 0 |  |  |  |
  Thyrotropin: Low (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Thyrotropin: Low (at baseline) to Missing (at post baseline) |  | 0 |  |  |  |
  Thyrotropin: Normal (at baseline) to Low (at post baseline): number analyzed (Participants) | 6 | 4 | 5 | 18 | 22 | 10
  Thyrotropin: Normal (at baseline) to Low (at post baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Thyrotropin: Normal (at baseline) to Normal (at post baseline): number analyzed (Participants) | 6 | 4 | 5 | 18 | 22 | 10
  Thyrotropin: Normal (at baseline) to Normal (at post baseline) | 2 | 4 | 5 | 14 | 12 | 5
  Thyrotropin: Normal (at baseline) to High (at post baseline): number analyzed (Participants) | 6 | 4 | 5 | 18 | 22 | 10
  Thyrotropin: Normal (at baseline) to High (at post baseline) | 3 | 0 | 0 | 4 | 5 | 5
  Thyrotropin: Normal (at baseline) to Missing (at post baseline): number analyzed (Participants) | 6 | 4 | 5 | 18 | 22 | 10
  Thyrotropin: Normal (at baseline) to Missing (at post baseline) | 1 | 0 | 0 | 0 | 5 | 0
  Thyrotropin: High (at baseline) to Low (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1 | 5 | 1
  Thyrotropin: High (at baseline) to Low (at post baseline) |  | 0 | 0 | 0 | 0 | 0
  Thyrotropin: High (at baseline) to Normal (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1 | 5 | 1
  Thyrotropin: High (at baseline) to Normal (at post baseline) |  | 0 | 1 | 0 | 0 | 1
  Thyrotropin: High (at baseline) to High (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1 | 5 | 1
  Thyrotropin: High (at baseline) to High (at post baseline) |  | 1 | 0 | 1 | 5 | 0
  Thyrotropin: High (at baseline) to Missing (at post baseline): number analyzed (Participants) | 0 | 1 | 2 | 1 | 5 | 1
  Thyrotropin: High (at baseline) to Missing (at post baseline) |  | 0 | 1 | 0 | 0 | 0

15. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Number of Participants With Clinically Significant Urinalysis Finding
Description: Urinalysis laboratory parameters/abnormalities: Decimal logarithm of reciprocal of hydrogen ion activity (pH), specific gravity, protein, glucose, ketones, nitrite, blood, leukocyte esterase, microscopy (if urine tested positive for blood or protein). Clinical significance was judged by investigator.
Time Frame: as for outcome 10
Population: Safety set included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Number of Participants With Newly Occurring Clinically Notable Vital Sign Abnormalities
Description: Vital signs included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate, body temperature and weight. Low SBP: less than or equal to (<=)90 millimeter of mercury (mmHg) with decrease from baseline of >=20 mmHg. High SBP: >=160 mmHg with increase from baseline of >=20 mmHg. Low DBP: <=50 mmHg with decrease from baseline of >=15 mmHg. High DBP: >=100 mmHg with increase from baseline of >=15 mmHg. Low heart rate: <=50 beats/min with decrease from baseline of >=15 beats/min. High heart rate: >=120 beats/min with increase from baseline of >=15 beats/min. Low temperature: <=36 degree Celsius (C). High temperature: >=37.5 degree C. Low Weight: decrease from baseline >=20%. High weight: increase from baseline >=10%.
Time Frame: as for outcome 10
Population: Safety set included all participants who received at least 1 dose (partial or full) of ARRY-382 or pembrolizumab. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
Participants
  SBP: High: number analyzed (Participants) | 6 | 6 | 5 | 19 | 23 | 8
  SBP: High | 3 | 0 | 0 | 1 | 2 | 1
  SBP: Low: number analyzed (Participants) | 6 | 6 | 6 | 18 | 23 | 11
  SBP: Low | 1 | 0 | 0 | 0 | 1 | 0
  DBP: High: number analyzed (Participants) | 6 | 6 | 6 | 19 | 23 | 11
  DBP: High | 0 | 0 | 1 | 1 | 0 | 0
  DBP: Low: number analyzed (Participants) | 6 | 6 | 6 | 19 | 23 | 11
  DBP: Low | 1 | 0 | 0 | 0 | 1 | 0
  Heart Rate: High: number analyzed (Participants) | 6 | 6 | 6 | 19 | 21 | 11
  Heart Rate: High | 0 | 1 | 2 | 2 | 2 | 0
  Heart Rate: Low: number analyzed (Participants) | 6 | 6 | 6 | 19 | 23 | 11
  Heart Rate: Low | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: High: number analyzed (Participants) | 6 | 6 | 5 | 19 | 22 | 11
  Temperature: High | 1 | 0 | 1 | 1 | 3 | 1
  Temperature: Low: number analyzed (Participants) | 6 | 5 | 4 | 17 | 20 | 11
  Temperature: Low | 4 | 1 | 2 | 3 | 5 | 1
  Weight: High: number analyzed (Participants) | 5 | 6 | 6 | 19 | 22 | 11
  Weight: High | 1 | 0 | 0 | 0 | 2 | 0
  Weight: Low: number analyzed (Participants) | 5 | 6 | 6 | 19 | 22 | 11
  Weight: Low | 0 | 0 | 0 | 0 | 1 | 0

17. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Plasma Concentration Versus Time Profile of ARRY-382
Description: The lower limit of quantitation (LLOQ) for analyte ARRY-382 was 5.00 nanogram per milliliter (ng/mL).
Time Frame: Pre dose of ARRY-382 (120 minutes prior to administration): on Day 15 of Cycle 1, on Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9 , 10; 1 hour(hr) (±5 min), 2 hours(hrs) (±10 min), 4 hrs (±20 min) and 8 hrs (±30 min) post dose of ARRY-382 on Day 1 of Cycle 1, 2
Population: Pharmacokinetic (PK) set included all participants who had received any active study intervention (ARRY-382), with at least one post dose blood draw to determine plasma concentration of ARRY-382. Here "Number Analyzed" signifies number of participants evaluated for given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
nanogram per milliliter
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 6 | 5 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose | 283 (422) | 49.7 (1130) | 305 (263) | 664 (194) | 373 (282) | 695 (145)
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose | 542 (78.8) | 497 (201) | 827 (64.2) | 1060 (65.8) | 982 (101) | 1160 (57.2)
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose | 530 (37.9) | 845 (49.0) | 1130 (50.0) | 1010 (44.7) | 976 (72.6) | 937 (54.5)
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 8
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose | 384 (26.3) | 566 (28.8) | 757 (46.8) | 683 (43.7) | 662 (76.7) | 500 (52.6)
  Cycle 1 Day 15 / Pre ARRY-382 dose: number analyzed (Participants) | 5 | 3 | 2 | 10 | 16 | 7
  Cycle 1 Day 15 / Pre ARRY-382 dose | 616 (43.0) | 533 (34.2) | 888 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 862 (57.3) | 918 (79.1) | 485 (117)
  Cycle 2 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 2 | 6 | 3 | 5
  Cycle 2 Day 1 / Pre ARRY-382 dose | 576 (59.5) | 762 (6.44) | 1040 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 330 (2050) | 1550 (18.8) | 438 (86.5)
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 4 | 2 | 3 | 5 | 3 | 5
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose | 1170 (76.5) | 1310 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 1430 (195) | 1320 (97.5) | 2000 (14.3) | 1220 (64.2)
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 4
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose | 1530 (45.2) | 1600 (106) | 2560 (117) | 1830 (92.2) | 3000 (9.01) | 1580 (79.6)
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose | 1200 (57.6) | 2030 (35.1) | 2120 (126) | 1630 (66.6) | 2900 (4.73) | 1450 (62.7)
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose | 1100 (35.7) | 1680 (8.22) | 1440 (142) | 1530 (52.3) | 2150 (7.22) | 973 (75.5)
  Cycle 3 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 3 | 1 | 0 | 4 | 5 | 2
  Cycle 3 Day 1 / Pre ARRY-382 dose | 565 (39.5) | 305 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 554 (70.3) | 324 (391) | 336 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3.
  Cycle 4 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 2 | 0 | 0 | 4 | 4 | 1
  Cycle 4 Day 1 / Pre ARRY-382 dose | 405 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. |  |  | 1080 (119) | 728 (85.2) | 522 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 5 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 1 | 0 | 0 | 3 | 3 | 1
  Cycle 5 Day 1 / Pre ARRY-382 dose | NA (NA) — Since concentration was below quantifiable limit, geometric mean and geometric coefficient of variation could not be calculated. |  |  | 92.6 (13300) | 1000 (35.1) | 76.6 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 6 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 1
  Cycle 6 Day 1 / Pre ARRY-382 dose |  |  |  | 798 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. | 1100 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 518 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 7 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1
  Cycle 7 Day 1 / Pre ARRY-382 dose |  |  |  | 573 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 505 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 8 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 1 / Pre ARRY-382 dose |  |  |  | 424 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 9 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 9 Day 1 / Pre ARRY-382 dose |  |  |  | 350 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 10 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 10 Day 1 / Pre ARRY-382 dose |  |  |  | 244 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |

18. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Plasma Concentration Versus Time Profile of Metabolite AR00469099
Description: Drug ARRY-382 had its three metabolites AR00469099, AR00469100 and AR00470870. Plasma concentration of metabolite AR00469099 was reported in this outcome measure. The LLOQ for analyte AR00469099 was 1.00 ng/mL.
Time Frame: Pre dose of ARRY-382 (120 minutes prior to administration): on Day 15 of Cycle 1, on Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9 , 10; 1 hr (±5 min), 2 hrs (±10 min), 4 hrs (±20 min), and 8 hrs (±30 min) post dose of ARRY-382 on Day 1 of Cycle 1, 2
Population: PK set included all participants who had received any active study intervention (ARRY-382), with at least one post dose blood draw to determine plasma concentration of metabolite AR00469099. Here "Number Analyzed" signifies number of participants evaluated for given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
nanogram per milliliter
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 6 | 5 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose | 10.6 (750) | NA (NA) — Since concentration was below quantifiable limit, geometric mean and geometric coefficient of variation could not be calculated. | 8.57 (404) | 21.0 (234) | 7.95 (493) | 22.6 (164)
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose | 36.3 (219) | 19.6 (495) | 57.2 (151) | 66.2 (80.5) | 54.7 (177) | 60.8 (52.9)
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose | 69.5 (128) | 83.6 (69.2) | 170 (72.6) | 110 (48.9) | 113 (109) | 89.1 (39.5)
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 8
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose | 74.9 (85.3) | 96.4 (62.9) | 205 (88.7) | 119 (49.5) | 132 (101) | 75.7 (41.6)
  Cycle 1 Day 15 / Pre ARRY-382 dose: number analyzed (Participants) | 5 | 3 | 2 | 10 | 16 | 7
  Cycle 1 Day 15 / Pre ARRY-382 dose | 136 (30.8) | 73.7 (62.1) | 190 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 210 (78.8) | 250 (172) | 83.3 (132)
  Cycle 2 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 2 | 6 | 3 | 5
  Cycle 2 Day 1 / Pre ARRY-382 dose | 136 (67.7) | 199 (82.5) | 188 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 96.5 (2860) | 511 (189) | 77.1 (85.2)
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 4 | 2 | 3 | 5 | 3 | 5
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose | 133 (72.0) | 245 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 177 (94.7) | 254 (29.2) | 475 (173) | 102 (68.2)
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 4
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose | 166 (66.0) | 166 (133) | 241 (73.8) | 272 (36.2) | 510 (174) | 133 (54.1)
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose | 177 (89.6) | 208 (129) | 305 (62.0) | 298 (55.6) | 544 (168) | 157 (50.7)
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose | 210 (57.5) | 320 (71.9) | 313 (77.8) | 324 (44.1) | 561 (152) | 146 (58.5)
  Cycle 3 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 3 | 1 | 0 | 4 | 5 | 2
  Cycle 3 Day 1 / Pre ARRY-382 dose | 121 (81.8) | 31.0 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 123 (210) | 70.6 (243) | 54.0 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3.
  Cycle 4 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 2 | 0 | 0 | 4 | 4 | 1
  Cycle 4 Day 1 / Pre ARRY-382 dose | 79.9 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. |  |  | 157 (228) | 138 (30.0) | 70.3 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 5 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 1 | 0 | 0 | 3 | 3 | 1
  Cycle 5 Day 1 / Pre ARRY-382 dose | NA (NA) — Since concentration was below quantifiable limit, geometric mean and geometric coefficient of variation could not be calculated. |  |  | 11.5 (4020) | 170 (10.4) | 7.92 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 6 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 1
  Cycle 6 Day 1 / Pre ARRY-382 dose |  |  |  | 86.9 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. | 141 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 110 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 7 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1
  Cycle 7 Day 1 / Pre ARRY-382 dose |  |  |  | 61.5 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 103 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 8 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 1 / Pre ARRY-382 dose |  |  |  | 42.7 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 9 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 9 Day 1 / Pre ARRY-382 dose |  |  |  | 30.6 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 10 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 10 Day 1 / Pre ARRY-382 dose |  |  |  | 27.0 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |

19. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Plasma Concentration Versus Time Profile of Metabolite AR00469100
Description: Drug ARRY-382 had its three metabolites AR00469099, AR00469100 and AR00470870. Plasma concentration of metabolite AR00469100 was reported in this outcome measure. The LLOQ for analyte AR00469100 was 1.00 ng/mL.
Time Frame: as for outcome 18
Population: PK set included all participants who had received any active study intervention (ARRY-382), with at least one post dose blood draw to determine plasma concentration of metabolite AR00469100. Here "Number Analyzed" signifies number of participants evaluated for given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
nanogram per milliliter
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 6 | 5 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose | 19.5 (667) | NA (NA) — Since concentration was below quantifiable limit, geometric mean and geometric coefficient of variation could not be calculated. | 16.6 (584) | 61.0 (337) | 21.3 (553) | 75.4 (131)
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose | 47.1 (109) | 43.0 (468) | 71.0 (96.9) | 114 (69.1) | 81.9 (150) | 123 (51.2)
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose | 41.7 (79.2) | 82.7 (55.7) | 110 (40.5) | 102 (62.0) | 85.5 (84.8) | 101 (46.8)
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 8
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose | 28.2 (71.2) | 53.9 (42.5) | 67.7 (40.5) | 65.4 (64.8) | 56.4 (83.3) | 44.0 (50.5)
  Cycle 1 Day 15 / Pre ARRY-382 dose: number analyzed (Participants) | 5 | 3 | 2 | 10 | 16 | 7
  Cycle 1 Day 15 / Pre ARRY-382 dose | 70.7 (81.2) | 69.4 (24.5) | 116 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 106 (94.1) | 96.0 (85.3) | 60.8 (121)
  Cycle 2 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 2 | 6 | 3 | 5
  Cycle 2 Day 1 / Pre ARRY-382 dose | 60.1 (103) | 107 (45.5) | 146 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 35.2 (977) | 184 (91.1) | 57.1 (99.2)
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 4 | 2 | 3 | 5 | 3 | 5
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose | 105 (98.3) | 169 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 138 (228) | 116 (75.2) | 191 (92.5) | 173 (39.1)
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 4
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose | 138 (81.9) | 196 (81.9) | 268 (141) | 165 (81.7) | 265 (65.5) | 226 (66.5)
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose | 108 (108) | 228 (39.5) | 219 (131) | 139 (57.4) | 264 (75.1) | 164 (67.5)
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose | 104 (75.9) | 210 (27.1) | 161 (158) | 124 (39.5) | 218 (74.8) | 107 (77.8)
  Cycle 3 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 3 | 1 | 0 | 4 | 5 | 2
  Cycle 3 Day 1 / Pre ARRY-382 dose | 63.2 (108) | 57.3 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 73.2 (73.5) | 54.8 (255) | 32.7 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3.
  Cycle 4 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 2 | 0 | 0 | 4 | 4 | 1
  Cycle 4 Day 1 / Pre ARRY-382 dose | 31.1 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. |  |  | 108 (109) | 75.5 (88.7) | 67.6 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 5 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 1 | 0 | 0 | 3 | 3 | 1
  Cycle 5 Day 1 / Pre ARRY-382 dose | NA (NA) — Since concentration was below quantifiable limit, geometric mean and geometric coefficient of variation could not be calculated. |  |  | 14.0 (6560) | 112 (46.2) | 11.7 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 6 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 1
  Cycle 6 Day 1 / Pre ARRY-382 dose |  |  |  | 110 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. | 148 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 72.8 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 7 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1
  Cycle 7 Day 1 / Pre ARRY-382 dose |  |  |  | 73.2 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 67.4 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 8 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 1 / Pre ARRY-382 dose |  |  |  | 51.3 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 9 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 9 Day 1 / Pre ARRY-382 dose |  |  |  | 44.0 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 10 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 10 Day 1 / Pre ARRY-382 dose |  |  |  | 33.8 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |

20. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Plasma Concentration Versus Time Profile of Metabolite AR00470870
Description: Drug ARRY-382 had its three metabolites AR00469099, AR00469100 and AR00470870. Plasma concentration of metabolite AR00470870 was reported in this outcome measure. The LLOQ for analyte AR00470870 was 1.00 ng/mL.
Time Frame: as for outcome 18
Population: PK set included all participants who had received any active study intervention (ARRY-382), with at least one post dose blood draw to determine plasma concentration of metabolite AR00470870. Here "Number Analyzed" signifies number of participants evaluated for given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
nanogram per milliliter
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 6 | 5 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 1 hr Post ARRY-382 dose | 14.6 (835) | NA (NA) — Since concentration was below quantifiable limit, geometric mean and geometric coefficient of variation could not be calculated. | 11.7 (410) | 46.9 (403) | 12.6 (1100) | 71.7 (125)
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day 1 / 2 hrs Post ARRY-382 dose | 49.4 (193) | 36.7 (2940) | 68.7 (113) | 140 (97.9) | 74.8 (277) | 189 (59.5)
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 11
  Cycle 1 Day1 / 4 hrs Post ARRY-382 dose | 64.5 (101) | 159 (106) | 182 (73.7) | 191 (59.9) | 129 (116) | 220 (46.9)
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 6 | 6 | 7 | 17 | 26 | 8
  Cycle 1 Day1 / 8 hrs Post ARRY-382 dose | 53.7 (78.4) | 144 (71.3) | 162 (52.6) | 150 (56.8) | 123 (90.1) | 148 (46.7)
  Cycle 1 Day 15 / Pre ARRY-382 dose: number analyzed (Participants) | 5 | 3 | 2 | 10 | 16 | 7
  Cycle 1 Day 15 / Pre ARRY-382 dose | 105 (86.9) | 255 (11.0) | 231 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 259 (49.3) | 307 (74.0) | 242 (33.5)
  Cycle 2 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 2 | 6 | 3 | 5
  Cycle 2 Day 1 / Pre ARRY-382 dose | 99.1 (80.8) | 294 (49.3) | 216 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 83.4 (2600) | 285 (58.4) | 224 (34.1)
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose: number analyzed (Participants) | 4 | 2 | 3 | 5 | 3 | 5
  Cycle 2 Day 1 / 1 hr Post ARRY-382 dose | 122 (63.9) | 377 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 206 (68.5) | 244 (58.1) | 279 (53.8) | 316 (26.4)
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 4
  Cycle 2 Day 1 / 2 hrs Post ARRY-382 dose | 165 (49.3) | 444 (29.0) | 283 (68.8) | 337 (70.2) | 310 (47.2) | 462 (16.9)
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 4 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 4 hrs Post ARRY-382 dose | 149 (54.4) | 503 (26.8) | 327 (61.2) | 320 (65.9) | 348 (40.3) | 486 (18.9)
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose: number analyzed (Participants) | 4 | 3 | 3 | 6 | 3 | 5
  Cycle 2 Day 1 / 8 hrs Post ARRY-382 dose | 151 (58.9) | 460 (37.6) | 306 (47.9) | 337 (55.3) | 345 (36.1) | 401 (19.2)
  Cycle 3 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 3 | 1 | 0 | 4 | 5 | 2
  Cycle 3 Day 1 / Pre ARRY-382 dose | 118 (88.7) | 250 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 156 (87.0) | 194 (65.0) | 194 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3.
  Cycle 4 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 2 | 0 | 0 | 4 | 4 | 1
  Cycle 4 Day 1 / Pre ARRY-382 dose | 77.4 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. |  |  | 161 (113) | 263 (13.5) | 158 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 5 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 1 | 0 | 0 | 3 | 3 | 1
  Cycle 5 Day 1 / Pre ARRY-382 dose | NA (NA) — Since concentration was below quantifiable limit, geometric mean and geometric coefficient of variation could not be calculated. |  |  | 16.4 (10600) | 268 (18.2) | 33.8 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 6 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 1
  Cycle 6 Day 1 / Pre ARRY-382 dose |  |  |  | 73.5 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. | 419 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 192 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 7 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1
  Cycle 7 Day 1 / Pre ARRY-382 dose |  |  |  | 60.7 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  | 236 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated.
  Cycle 8 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 8 Day 1 / Pre ARRY-382 dose |  |  |  | 62.8 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 9 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 9 Day 1 / Pre ARRY-382 dose |  |  |  | 73.8 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |
  Cycle 10 Day 1 / Pre ARRY-382 dose: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 10 Day 1 / Pre ARRY-382 dose |  |  |  | 90.6 (NA) — Due to insufficient number of participants with events, geometric coefficient of variation could not be calculated. |  |

21. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Area Under the Plasma Concentration-Time Curve Over a Dosing Interval at Steady-State (AUCtau, ss) for ARRY-382 and Metabolites (AR00469099, AR00469100, and AR00470870)
Description: AUCtau was defined as area under the plasma concentration-time curve over the dosing interval, where dosing interval was 24 hours.
Time Frame: 0 to 24 hrs after administration of ARRY-382 on Day 1 of Cycle 2
Population: PK set included all participants who had received any active study intervention (ARRY-382), with at least one post dose blood draw to determine plasma concentration of ARRY-382 and its metabolites (AR00469099, AR00469100 and AR00470870). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 4 | 5
hour*nanogram per milliliter
  ARRY-382 | 22800 (44.2) | 30600 (26.6) | 30800 (130) | 32100 (65.7) | 47100 (10.2) | 20700 (70.6)
  AR00469099 | 4150 (63.5) | 4530 (106) | 5880 (78.8) | 7920 (18.9) | 14200 (123) | 2840 (61.8)
  AR00469100 | 2170 (85.9) | 3860 (33.9) | 3510 (142) | 2670 (53.4) | 5360 (62.8) | 2480 (73.9)
  AR00470870 | 3180 (59.0) | 9810 (29.3) | 6200 (45.2) | 6850 (61.2) | 7940 (36.9) | 8220 (20.3)

22. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Maximum Observed Plasma Concentration (Cmax) for ARRY-382 and Metabolites (AR00469099, AR00469100, and AR00470870)
Description: Cmax was obtained from plasma concentration time curve. Cmax at single dose was reported at Cycle1 Day 1 and Cmax at steady state was reported at Cycle 2 Day 1.
Time Frame: Pre dose of ARRY-382 (120 minutes prior to administration), 1 hr (±5 min), 2 hrs (±10 min), 4 hrs (±20 min), and 8 hrs (±30 min) after administration of ARRY-382 on Day 1 of Cycle 1 and 2
Population: PK set included all participants who had received any active study intervention (ARRY-382), with at least one post dose blood draw to determine plasma concentration of ARRY-382 and its metabolites (AR00469099, AR00469100 and AR00470870). Here "Number Analyzed" signifies number of participants evaluated for given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
nanogram per milliliter
  Cycle 1 Day 1 ARRY-382: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 ARRY-382 | 773 (60.2) | 995 (68.9) | 1330 (39.6) | 1240 (62.1) | 1290 (75.6) | 1260 (53.9)
  Cycle 2 Day 1 ARRY-382: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 ARRY-382 | 1560 (41.3) | 2260 (36.6) | 2560 (117) | 2130 (60.4) | 2820 (15.1) | 1580 (64.8)
  Cycle 1 Day 1 AR00469099: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469099 | 84.0 (102) | 100 (59.8) | 219 (83.8) | 119 (50.9) | 142 (97.9) | 95.4 (43.2)
  Cycle 2 Day 1 AR00469099: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00469099 | 212 (57.3) | 241 (103) | 328 (75.6) | 328 (44.0) | 646 (111) | 161 (50.8)
  Cycle 1 Day 1 AR00469100: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469100 | 61.2 (78.3) | 104 (86.5) | 122 (41.7) | 132 (70.0) | 116 (98.3) | 138 (46.5)
  Cycle 2 Day 1 AR00469100: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00469100 | 138 (81.6) | 257 (36.4) | 268 (141) | 181 (56.9) | 279 (54.9) | 215 (52.5)
  Cycle 1 Day 1 AR00470870: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00470870 | 70.1 (95.1) | 174 (92.5) | 196 (58.5) | 193 (60.5) | 147 (98.9) | 231 (50.8)
  Cycle 2 Day 1 AR00470870: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00470870 | 172 (51.6) | 534 (22.0) | 333 (60.7) | 373 (60.6) | 363 (30.9) | 486 (18.9)

23. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Ctrough at Steady State for ARRY-382 and Metabolites (AR00469099, AR00469100, and AR00470870)
Description: Measured concentration at the pre-dose at steady-state.
Time Frame: Pre dose of ARRY-382 (120 minutes prior to administration) on Day 1 of Cycle 2
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 4 | 5
nanogram per milliliter
  ARRY-382 | 576 (59.5) | 667 (27.7) | 627 (126) | 878 (70.1) | 1480 (17.5) | 438 (86.5)
  AR00469099 | 136 (67.7) | 146 (105) | 161 (105) | 277 (27.1) | 557 (136) | 77.1 (85.2)
  AR00469100 | 60.1 (103) | 96.0 (43.9) | 83.6 (137) | 82.4 (57.1) | 193 (71.3) | 57.1 (99.2)
  AR00470870 | 99.1 (80.8) | 313 (41.7) | 185 (27.9) | 232 (58.5) | 302 (48.1) | 224 (34.1)

24. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Time to Reach Maximum Observed Plasma Concentration (Tmax) for ARRY-382 and Metabolites (AR00469099, AR00469100, and AR00470870)
Description: Tmax was obtained from plasma concentration time curve. Tmax at single dose was reported at Cycle 1 Day 1 and Tmax at steady state was reported at Cycle 2 Day 1.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
hours
  Cycle 1 Day 1 ARRY-382: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 ARRY-382 | 2.00 [1.00 to 7.95] | 4.01 [1.25 to 4.05] | 4.07 [0.983 to 8.00] | 1.97 [0.950 to 4.17] | 2.00 [0.967 to 8.00] | 2.00 [1.00 to 4.10]
  Cycle 2 Day 1 ARRY-382: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 ARRY-382 | 2.00 [2.00 to 7.95] | 4.18 [1.85 to 7.48] | 1.98 [1.97 to 2.00] | 2.00 [1.00 to 7.50] | 3.03 [2.00 to 4.08] | 2.00 [1.83 to 4.17]
  Cycle 1 Day 1 AR00469099: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469099 | 7.98 [4.00 to 8.02] | 7.81 [3.97 to 8.00] | 7.95 [4.00 to 8.02] | 5.88 [3.98 to 8.00] | 5.83 [1.92 to 8.03] | 4.17 [2.00 to 8.00]
  Cycle 2 Day 1 AR00469099: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00469099 | 7.94 [4.10 to 8.05] | 7.68 [3.85 to 8.00] | 8.00 [4.00 to 8.00] | 7.50 [4.00 to 8.00] | 5.90 [0.00 to 8.00] | 4.05 [2.00 to 7.50]
  Cycle 1 Day 1 AR00469100: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469100 | 2.00 [1.00 to 4.07] | 2.98 [1.25 to 4.05] | 4.07 [0.983 to 8.00] | 2.00 [1.00 to 4.17] | 2.00 [0.967 to 8.02] | 2.00 [1.00 to 4.10]
  Cycle 2 Day 1 AR00469100: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00469100 | 2.00 [2.00 to 7.95] | 3.03 [1.85 to 7.48] | 1.98 [1.97 to 2.00] | 1.98 [1.00 to 7.50] | 3.90 [2.00 to 4.03] | 2.00 [0.917 to 3.75]
  Cycle 1 Day 1 AR00470870: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00470870 | 3.00 [2.00 to 8.02] | 4.03 [1.83 to 8.00] | 4.07 [4.00 to 8.00] | 4.00 [2.00 to 7.58] | 4.07 [1.92 to 8.02] | 3.80 [1.88 to 4.15]
  Cycle 2 Day 1 AR00470870: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00470870 | 3.00 [2.00 to 7.95] | 4.18 [1.85 to 7.48] | 8.00 [4.00 to 8.00] | 4.03 [1.95 to 7.50] | 5.78 [4.00 to 8.00] | 4.05 [3.75 to 4.17]

25. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Metabolite-to-Parent Ratio (MR) for ARRY-382 and Metabolites (AR00469099, AR00469100, and AR00470870)
Description: Different MR reported for single dose calculated at Cycle 1 Day 1 were as follows: 1) MRAUClast = ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight, where AUClast was area under the plasma concentration-time curve from zero to the last measurable time point; 2) MRCmax = ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight. Different MR reported for steady state calculated at Cycle 2 Day 1 were as follows: 1) MRAUCtau,ss = ratio of AUCtau,ss values of the metabolite compared to parent, corrected for molecular weight, where AUCtau was area under the plasma concentration-time curve over a dosing interval at steady-state; 2) MRCmax,ss = Ratio of Cmax,ss values of the metabolite compared to parent, corrected for molecular weight.
Time Frame: Pre dose of ARRY-382 (120 minutes prior to administration),1 hrs (±5 min), 2 hrs (±10 min), 4 hrs (±20 min), and 8 hrs (±30 min) after administration of ARRY-382 on Day 1 of Cycle 1 and 2
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 6 | 6 | 7 | 19 | 27 | 11
ratio
  Cycle 1 Day 1 AR00469099 MRAUClast: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469099 MRAUClast | 0.115 (86.8) | 0.101 (47.9) | 0.151 (70.9) | 0.101 (45.7) | 0.108 (63.4) | 0.0821 (31.3)
  Cycle 1 Day 1 AR00469099 MRCmax: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469099 MRCmax | 0.106 (58.8) | 0.0979 (74.9) | 0.160 (79.5) | 0.0929 (46.5) | 0.107 (71.8) | 0.0734 (38.3)
  Cycle 2 Day 1 AR00469099 MRAUCtau,ss: number analyzed (Participants) | 4 | 4 | 3 | 5 | 4 | 5
  Cycle 2 Day 1 AR00469099 MRAUCtau,ss | 0.177 (35.6) | 0.144 (80.3) | 0.186 (84.6) | 0.240 (69.0) | 0.292 (132) | 0.134 (27.5)
  Cycle 2 Day 1 AR00469099 MRCmax,ss: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00469099 MRCmax,ss | 0.132 (20.5) | 0.103 (68.2) | 0.125 (74.8) | 0.150 (89.9) | 0.222 (108) | 0.0991 (24.0)
  Cycle 1 Day 1 AR00469100 MRAUClast: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469100 MRAUClast | 0.0817 (40.7) | 0.101 (33.4) | 0.0934 (31.0) | 0.104 (39.3) | 0.0883 (41.2) | 0.108 (22.9)
  Cycle 1 Day 1 AR00469100 MRCmax: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00469100 MRCmax | 0.0811 (45.0) | 0.107 (35.0) | 0.0941 (21.8) | 0.109 (47.2) | 0.0923 (41.3) | 0.112 (29.8)
  Cycle 2 Day 1 AR00469100 MRAUCtau,ss: number analyzed (Participants) | 4 | 4 | 3 | 5 | 4 | 5
  Cycle 2 Day 1 AR00469100 MRAUCtau,ss | 0.0978 (43.8) | 0.129 (27.1) | 0.117 (13.1) | 0.0853 (13.8) | 0.117 (66.4) | 0.123 (40.8)
  Cycle 2 Day 1 AR00469100 MRCmax,ss: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00469100 MRCmax,ss | 0.0909 (41.4) | 0.116 (29.3) | 0.108 (24.5) | 0.0873 (19.2) | 0.101 (52.8) | 0.140 (44.3)
  Cycle 1 Day 1 AR00470870 MRAUClast: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00470870 MRAUClast | 0.0946 (104) | 0.159 (42.7) | 0.127 (44.9) | 0.151 (71.1) | 0.106 (64.0) | 0.176 (72.4)
  Cycle 1 Day 1 AR00470870 MRCmax: number analyzed (Participants) | 6 | 6 | 7 | 18 | 26 | 11
  Cycle 1 Day 1 AR00470870 MRCmax | 0.0775 (119) | 0.149 (26.6) | 0.126 (30.4) | 0.133 (78.0) | 0.0974 (51.4) | 0.156 (71.6)
  Cycle 2 Day 1 AR00470870 MRAUCtau,ss: number analyzed (Participants) | 4 | 4 | 3 | 5 | 4 | 5
  Cycle 2 Day 1 AR00470870 MRAUCtau,ss | 0.119 (80.2) | 0.273 (43.1) | 0.172 (66.7) | 0.182 (69.3) | 0.144 (41.1) | 0.340 (59.0)
  Cycle 2 Day 1 AR00470870 MRCmax,ss: number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
  Cycle 2 Day 1 AR00470870 MRCmax,ss | 0.0941 (84.4) | 0.201 (36.1) | 0.111 (42.7) | 0.150 (66.6) | 0.110 (31.3) | 0.263 (59.6)

26. Secondary Outcome: Phase 1b, Part A and Phase 2 Cohorts: Accumulation Ratio (R) for ARRY-382 and Metabolites (AR00469099, AR00469100, and AR00470870)
Description: Accumulation ratio was calculated and reported for Cmax as RCmax and for AUC as RAUC. RCmax = Cmax at steady-state on Day 1 of Cycle 2 divided by Cmax on Day 1 of Cycle 1. RAUC = AUC from zero to 8 hours after drug administration at steady-state on Day 1 of Cycle 2 divided by AUC from zero to 8 hours after drug administration on Day 1 of Cycle 1.
Time Frame: Pre dose of ARRY-382 (120 minutes prior to administration),1 hr (±5 min), 2 hrs (±10 min), 4 hrs (±20 min), and 8 hrs (±30 min) after administration of ARRY-382 on Day 1 of Cycle 1 and 2
Population: PK set included all participants who had received any active study intervention (ARRY-382), with at least one postdose blood draw to determineplasma concentration of ARRY-382 and its metabolites (AR00469099, AR00469100 and AR00470870). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
Number analyzed (Participants) | 4 | 4 | 3 | 6 | 4 | 5
ratio
  Cycle 2 Day 1 ARRY-382 RAUC: number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 4
  Cycle 2 Day 1 ARRY-382 RAUC | 3.03 (47.9) | 1.92 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 3.52 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 2.67 (36.2) | 3.41 (23.6) | 1.87 (16.7)
  Cycle 2 Day 1 ARRY-382 RCmax | 2.53 (48.2) | 2.51 (95.7) | 2.28 (54.2) | 2.52 (39.9) | 2.07 (53.6) | 1.62 (24.7)
  Cycle 2 Day 1 AR00469099 RAUC: number analyzed (Participants) | 3 | 1 | 2 | 2 | 3 | 4
  Cycle 2 Day 1 AR00469099 RAUC | 4.03 (93.0) | 4.36 (NA) — Since only 1 evaluable participant, geometric coefficient of variation could not be calculated. | 4.28 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 4.67 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 4.95 (41.8) | 2.07 (23.8)
  Cycle 2 Day 1 AR00469099 RCmax | 3.03 (53.4) | 2.54 (52.0) | 2.47 (38.5) | 3.19 (36.7) | 3.56 (48.4) | 1.93 (37.4)
  Cycle 2 Day 1 AR00469100 RCmax | 2.67 (46.1) | 2.60 (157) | 2.50 (65.1) | 2.44 (41.3) | 2.08 (49.0) | 1.76 (29.5)
  Cycle 2 Day 1 AR00469100 RAUC: number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 4
  Cycle 2 Day 1 AR00469100 RAUC | 3.49 (51.7) | 1.97 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 3.96 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 2.64 (36.3) | 3.84 (13.5) | 1.93 (23.0)
  Cycle 2 Day 1 AR00470870 RAUC: number analyzed (Participants) | 3 | 1 | 2 | 2 | 3 | 4
  Cycle 2 Day 1 AR00470870 RAUC | 3.47 (94.9) | 4.48 (NA) — Since only 1 evaluable participant, geometric coefficient of variation could not be calculated. | 2.73 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 4.01 (NA) — As planned geometric coefficient of variation would not be calculated and reported if evaluable participants were less than 3. | 3.30 (61.9) | 2.03 (23.9)
  Cycle 2 Day 1 AR00470870 RCmax | 2.72 (54.5) | 3.59 (95.3) | 2.02 (20.1) | 2.39 (48.6) | 2.03 (38.7) | 1.77 (31.0)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study treatment (for Phase 1b: maximum up to 34.7 months, for Phase 2: maximum up to 13.5 months)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety set was evaluated.
Arm/Group | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 1b, Part B: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2, Part C: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort
All-Cause Mortality (participants affected / at risk) | 4/6 | 6/6 | 5/7 | 1/1 | 1/2 | 10/19 | 20/27 | 5/11
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 3/7 | 1/1 | 1/2 | 8/19 | 15/27 | 5/11
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/7 | 1/1 | 2/2 | 19/19 | 26/27 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=6) | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=6) | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=7) | Phase 1b, Part B: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=1) | Phase 2, Part C: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=2) | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort (N=19) | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort (N=27) | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Part A: 200 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=6) | Phase 1b, Part A: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=6) | Phase 1b, Part A: 400 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=7) | Phase 1b, Part B: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=1) | Phase 2, Part C: 300 mg ARRY-382 + 2 mg/kg Pembrolizumab (N=2) | Phase 2: PD-1/PD-L1 Inhibitor-Refractory Cohort (N=19) | Phase 2: Pancreatic Ductal Adenocarcinoma (PDA) Cohort (N=27) | Phase 2: Platinum-resistant Ovarian Cancer (prOVCA) Cohort (N=11)
Aspartate aminotransferase increased (Investigations) | 2 | 6 | 4 | 0 | 0 | 8 | 9 | 4
Blood creatine phosphokinase increased (Investigations) | 2 | 3 | 3 | 0 | 0 | 9 | 5 | 2
Alanine aminotransferase increased (Investigations) | 2 | 3 | 2 | 0 | 0 | 3 | 5 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 3 | 0 | 0 | 5 | 4 | 0
Lipase increased (Investigations) | 1 | 4 | 1 | 0 | 0 | 6 | 1 | 0
Amylase increased (Investigations) | 1 | 3 | 1 | 0 | 0 | 4 | 2 | 0
Weight decreased (Investigations) | 1 | 0 | 2 | 0 | 0 | 3 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aldolase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 3 | 0 | 1 | 10 | 16 | 3
Pyrexia (General disorders) | 2 | 1 | 2 | 0 | 0 | 2 | 1 | 3
Chills (General disorders) | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 0 | 9 | 12 | 5
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 8 | 9 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 4 | 6 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric varices (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 0 | 0 | 5 | 9 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 5 | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 3 | 9 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thyroiditis acute (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 8 | 4 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgraphia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT02880371/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT02880371/SAP_001.pdf